CLINICAL TRIAL: NCT03297853
Title: Prevalence, Management and Follow-up of Patients With Addiction to Opioid Analgesics
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0305
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2017-09

CONDITIONS: Analgesics Grade 2's Addiction
Keywords: Descriptive; Support; Retrospective; survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The demand for addiction care for patients with addiction to analgesics increases with the number of prescription of analgesics grade 2; this is a public health problem There is no support for repositories to date in the context of addiction analgesics grade 2.

Risk factors of misuse as well as diagnostic tools were identified.

DETAILED DESCRIPTION:
The demand for addiction care for patients with addiction to analgesics increases with the number of prescription of analgesics grade 2; this is a public health problem There is no support for repositories to date in the context of addiction analgesics grade 2.

Risk factors of misuse as well as diagnostic tools were identified. The objectives of our research are to determine the characteristics of the individuals suffering from an addiction to analgesics of level 2 followed in consultation of addictology in the hospital of Montpellier and Nimes and to describe the type of follow-up proposed to the patients in these two centers. It is a retrospective and descriptive study.

As part of this research, we will solicit all the patients followed in consultation of addictology or in hospitalization to the hospital of Montpellier or Nîmes for an addiction to the analgesics of grade 2 between the 1st of January 2014 and the 10th of July 2017 with requests of management for withdrawal or reduction of doses, opioid analgesics in the absence of pain or in chronic non-cancer pain, opioid analgesics to avoid withdrawal syndrome or hyperalgesia and consumptions chronic to dosages inadequate to the functional complaint evaluated by the rhumatology or algology services.

The data are collected in the medical file at the two participating institutions (Montpellier and Nîmes) and if necessary, patients not seen in consultation for more than 6 months will be recontacted.

ELIGIBILITY:
Inclusion Criteria:

* Requests for management for weaning or reduction of doses
* Take opioid analgesics in the absence of pain or as part of chronic non-cancer pain
* Opioid analgesics to prevent withdrawal syndrome or hyperalgesia
* Chronic consumption at inadequate dosages compared to the functional complaint evaluated by the MPR / Algologie services
* Patients over 18 years and who agree with the study

Exclusion criteria:

* language barrier
* severe cognitive and / or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending addictology or hospitalization in Montpellier or Nîmes for an addiction to analgesics grade 2 between the 1st ofJanuary 2014 and the 22th of january 2017
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
50/5000 Prevalence of demand for care in addictology | 1 day
  Prevalence of demand for addictive care in subjects with addiction to analgesics in level 2

SECONDARY OUTCOMES:
Types of support proposed | 1 day
  Types of support proposed
Assessment of analgesic dependence | 1 day
  Assessment of analgesic dependence
History of analgesic use | 1 day
  History of analgesic use
quality of life | 1 day
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: TARUFFI Floriane, Doctor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC